CLINICAL TRIAL: NCT03455309
Title: A Phase 2 Double-blind Placebo-controlled Study to Evaluate the Safety, Immunogenicity and Efficacy of NDV-3A Vaccine in Preventing S. Aureus Colonization
Brief Title: Evaluation of NDV-3A Vaccine in Preventing S. Aureus Colonization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaDigm Therapeutics, Inc. (Industry)
Collaborators: Infectious Diseases Clinical Research Program (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NDV3A-006; IDCRP-104 (Other: IDCRP, USU)
Record Dates: First submitted 2018-02-13; First posted 2018-03-06 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Staphylococcus Aureus
Keywords: Als3; SSTI; vaccine; NDV-3A; incident nasal colonization
MeSH Terms: conditions — Staphylococcal Infections; Amyotrophic Lateral Sclerosis 3

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled, randomized study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor, principal investigator and study site are all blinded but can access key if safety issues require unblinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NDV-3A (Active Comparator): 0.5 mL dose containing 300 micrograms of recombinant Als3 protein in phosphate-buffered saline and 0.5 mg aluminum as aluminum hydroxide
  Interventions: Biological: NDV-3A
- Placebo (Placebo Comparator): 0.5 mL dose containing phosphate-buffered saline and 0.5 mg aluminum as aluminum hydroxide
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NDV-3A — Single dose administered by intramuscular injection
  Arms: NDV-3A
Biological: Placebo — Single dose administered by intramuscular injection
  Arms: Placebo

SUMMARY:
The proposed study aims to further evaluate the safety and immunogenicity of a candidate S. aureus vaccine NDV-3A, as well as its efficacy against acquisition of S. aureus

DETAILED DESCRIPTION:
The investigators will conduct a Phase 2 clinical trial to evaluate the safety, immunogenicity, and efficacy of candidate vaccine NDV-3A (NovaDigm Therapeutics, Inc.) to prevent incident nasal acquisition of S. aureus among a population of military recruits at increased risk for S. aureus colonization and disease. Colonization is a risk factor for skin and soft tissue infection (SSTI), and the anterior nares is an important reservoir for S. aureus. Use of S. aureus nasal colonization (specifically, incident nasal colonization with S. aureus post-vaccination) as a primary endpoint will allow the investigators to pursue a statistically-valid and meaningful parameter related to S. aureus SSTI. The proposed trial may yield evidence to warrant evaluation of NDV-3A efficacy against SSTI in a large-scale, Phase 2/3 trial in this high risk population.

ELIGIBILITY:
Inclusion Criteria:

* Active duty, male subject, 17-35 years of age, inclusive, at the time of screening.
* Assigned to one of the selected companies/battalions
* Informed of the nature of the study and has agreed to and is able to read, review, and sign the informed consent document prior to screening.
* Free of known significant health problems as established by the requirements to be enrolled in a military training program before entering into the study.
* Agrees to be reachable by phone, email or letter at 6 months post-vaccination.

Exclusion Criteria:

* Reports receiving any investigational drug, investigational vaccine, or investigational device within 30 days prior to dosing; subjects will be allowed to receive routine vaccinations associated with training and any other prescribed medications not in the exclusion criteria.
* Presence of clinically significant SSTI (e.g., cellulitis, abscess) at screening or other skin or skin structure infections that would confound the interpretation of clinical response.
* Reports a history of allergic response(s), anaphylaxis, or other serious reactions to previous vaccinations.
* Reports a history of allergies to yeast
* Reports a history of anaphylaxis or other serious reactions to aluminum.
* Reports a history of autoimmune disease (psoriasis, etc.)
* Seropositive for HIV antibody.
* Reports the use of any immunosuppressive drugs, including systemic corticosteroids (more than 14 days at a dose of >20 mg/day prednisone or equivalent), within 4 weeks prior to dosing.
* Reports receiving any blood products within 3 months prior to dosing.
* Reports donating blood/plasma within 28 days prior to dosing.
* Illness causing temperature ≥ 100.4°F
* Evidence of abnormal, unresolved laboratory results in the subject's medical record for the following tests: hemoglobin, white blood cell count, platelet count, creatinine, and alanine aminotransferase
* Any other medical and/or social reason which, in the opinion of the investigator(s), would increase the subject's risk of having an adverse reaction as a result of participation in the study.

Ages: 17 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 382 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Prevent acquisition of incident Staphylococcus aureus nasal colonization | 56 days post-vaccination
  Change in incident Staphylococcus aureus nasal colonization by study day 56 in a population of US Army trainees at Ft. Benning, GA

SECONDARY OUTCOMES:
Evaluation of the efficacy of the NDV-3A vaccine | 0-90 days
  Describe SSTI rates within the training company as defined by the development of skin and soft tissue infection (SSTI) over the training period as compared to other companies in the battalion as well as historical data
Evaluation of the efficacy of the NDV-3A vaccine | 0-90 days
  Describe NDV-3A-associated delay in time to first nasal acquisition of S. aureus colonization
Evaluation of the efficacy of the NDV-3A vaccine | 0-90 days
  Describe reduction in cross-sectional prevalence of S. aureus nasal/oral colonization
Evaluation of safety and tolerability in all subjects | 0-7 days
  Occurrence of solicited adverse events (AE) over a 7-day follow-up period following vaccination
Evaluation of safety and tolerability in all subjects | 0-28 days
  Occurrence of unsolicited AEs over a 28-day follow-up period following vaccination
Evaluation of safety and tolerability in all subjects | 0-90 days
  Occurrence of serious adverse events (SAE) or Adverse Events of Special Interest (AESI) at any time during the study period (enrollment to final in-person follow-up visit)
Measurement and characterization of immunogenicity of NDV-3A | 0-90 days
  Describe the humoral immune response induced by NDV-3A using ELISA analysis of serum
Measurement and characterization of immunogenicity of NDV-3A | 0-14 days
  Describe the cell mediated immune responses induced by NDV-3A using ELISpot analysis of PBMCs
Describe the impact of NDV-3A on S. aureus acquisition and transmission | 0-90 days
  Following determination of taxonomy (via sequencing of 16S rRNA), determine the relative abundance and distribution of, and change in, bacterial species colonizing the nose and throat (i.e. nasal/oral microbiome) of military trainees during the training period.
Describe the impact of NDV-3A on S. aureus acquisition and transmission | 0-90 days
  Compare the compositions of the nasal/oral microbiome between study groups to assess the impact of NDV-3A vaccine on the nasal/oral microbiome.
Describe the impact of NDV-3A on S. aureus acquisition and transmission | 0-90 days
  Utilize a combination of epidemiologic, microbiologic, and genomic data on colonization isolates to describe the intra-class transmission dynamics of S. aureus among congregate military trainees
Describe the impact of NDV-3A on S. aureus acquisition and transmission | 0-90 days
  Conduct whole genome sequencing on isolates to describe the intra- and inter-host concordance of infecting and colonizing strains of S. aureus

CONTACTS AND LOCATIONS:
Overall Officials: Jason W Bennett, MD, Principal Investigator — USU IDCRP
Locations (1):
- Fort Benning, Fort Benning, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeaman MR, Filler SG, Chaili S, Barr K, Wang H, Kupferwasser D, Hennessey JP Jr, Fu Y, Schmidt CS, Edwards JE Jr, Xiong YQ, Ibrahim AS. Mechanisms of NDV-3 vaccine efficacy in MRSA skin versus invasive infection. Proc Natl Acad Sci U S A. 2014 Dec 23;111(51):E5555-63. doi: 10.1073/pnas.1415610111. Epub 2014 Dec 8. PMID 25489065
- [Result] Schmidt CS, White CJ, Ibrahim AS, Filler SG, Fu Y, Yeaman MR, Edwards JE Jr, Hennessey JP Jr. NDV-3, a recombinant alum-adjuvanted vaccine for Candida and Staphylococcus aureus, is safe and immunogenic in healthy adults. Vaccine. 2012 Dec 14;30(52):7594-600. doi: 10.1016/j.vaccine.2012.10.038. Epub 2012 Oct 22. PMID 23099329